CLINICAL TRIAL: NCT06190119
Title: Comparative Analysis of Aqueous Humor Adipokines in Patients With Glaucoma and Healthy Controls
Brief Title: Comparison of Aqueous Humor Adipokines in Glaucoma Patients and Healthy Controls
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2023196
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Glaucoma; Adipokines
Keywords: Glaucoma；Adipokines；Neuroinflammation
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — aqueous humor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POAG Group: POAG patients who underwent filtering surgery, cataract surgery or MIGS.
  Interventions: Other: none intervention
- Control Group: Healthy patients who underwent cataract surgery.
  Interventions: Other: none intervention

INTERVENTIONS:
Other: none intervention — This study has no intervention

SUMMARY:
The purpose of this study is to observe whether there are differences in adipokines in the aqueous humor between patients with primary open-angle glaucoma (POAG) and healthy controls

DETAILED DESCRIPTION:
1. Inclusion criteria: Patients aged 18 years or older, diagnosed with primary open-angle glaucoma (POAG) and healthy controls (who underwent cataract surgery).

2. Exclusion criteria:

1. Other Ocular Diseases: Patients with concurrent ocular diseases such as macular degeneration, retinal detachment, etc., are excluded.
2. Ocular Surgery History: individuals who have undergone intraocular or laser surgery within the past 6 months, except for uncomplicated cataract surgery.
3. History of Ocular Trauma or Inflammation
4. Systemic Diseases or Mental Disorders: Patients with systemic diseases(e.g., diabetes, rheumatoid arthritis) and those with mental disorders are excluded.
5. Pregnancy or Lactation: Females who are pregnant or lactating are excluded.
6. Presence of any retinal or optic nerve disease other than glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, diagnosed with primary open-angle glaucoma (POAG) and healthy controls (who underwent cataract surgery).

Exclusion Criteria:

* Other Ocular Diseases: Patients with concurrent ocular diseases such as macular degeneration, retinal detachment, etc., are excluded.
* Ocular Surgery History: individuals who have undergone intraocular or laser surgery within the past 6 months, except for uncomplicated cataract surgery.
* History of Ocular Trauma or Inflammation
* Systemic Diseases or Mental Disorders: Patients with systemic diseases(e.g., diabetes, rheumatoid arthritis) and those with mental disorders are excluded.
* Pregnancy or Lactation: Females who are pregnant or lactating are excluded.
* Presence of any retinal or optic nerve disease other than glaucoma.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: POAG group and Control group are recruited from people who underwnt anti-glaucoma surgery and cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2023-10-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of adipokines in aqueous humor | Cross-sectional baseline
  Aqueous humor samples were assessed for adipokines and inflammatory cytokines by Luminex bead-based multiplex array

CONTACTS AND LOCATIONS:
Overall Officials: Chun Zhang, Ph.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hosipital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No